CLINICAL TRIAL: NCT03635684
Title: Evaluation of Efficacy and Safety of Subcutaneous Acetaminophen in Geriatrics and Palliative Care
Brief Title: Evaluation of Efficacy and Safety of Subcutaneous Acetaminophen
Acronym: APAPSubQ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Joe El Khoury, Principal Investigator, Saint-Joseph University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APAPSC2018
Record Dates: First submitted 2018-05-18; First posted 2018-08-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pain; Fever; Drug Effect; Drug Reaction
Keywords: Acetaminophen; Palliative Care; Infusions, Subcutaneous; Treatment Outcome; Geriatrics; Gerontology
MeSH Terms: conditions — Pain; Fever; Drug-Related Side Effects and Adverse Reactions | interventions — Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC Acetaminophen (Experimental): Palliative Care or Geriatric Patients who receive subcutaneous Acetaminophen for pain or fever relief
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Subcutaneous infusion of Acetaminophen over 20 to 30 minutes, with evaluation of:
  * local side effects;
  * pain and/or fever;
  at time of infusion, after 30 minutes, 60 minutes and 180 minutes.
  Other Names: Perfalgan; Paracetamol Macopharma

SUMMARY:
Subcutaneous perfusion is an underused technique, the effectiveness of which has been demonstrated.

A number of drugs of different therapeutic classes, including morphine, have a good level of scientific evidence for use by this route.

Subcutaneous Acetaminophen injection is being used in some medical centers, mainly in Europe, despite the lack of definite evidence on its efficacy.

This study aims to quantify the degree of effectiveness of subcutaneous Acetaminophen infusions for pain or fever in Geriatrics and Palliative Care, as well as determining its safety.

DETAILED DESCRIPTION:
Subcutaneous perfusion is an underused technique, the effectiveness of which has been demonstrated. It is mainly used in Palliative Care and Geriatrics when a venous line is not available. It is a simple and comfortable technique that allows to administer solutes and / or medications continuously or discontinuously in the subcutaneous tissue.

A number of drugs of different therapeutic classes, including morphine, have a good level of scientific evidence for use by this route.

Subcutaneous Acetaminophen injection is being used in some medical centers, mainly in Europe, despite the lack of definite evidence on its efficacy. It is sometimes accused of causing pain at the injection site; it seems that this is not the case if it is infused slowly, over 20 minutes to 30 minutes. There is no report of serious local effects.

The consultation palliative care team at Hôtel-Dieu de France (HDF) has used subcutaneous Acetaminophen infusions repeatedly without adverse effects since January 2014.

This study aims to quantify the degree of effectiveness of subcutaneous Acetaminophen infusions for pain or fever in Geriatrics and Palliative Care, as well as determining its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by the Palliative Care Consultation Team, patients admitted in the Palliative Care Unit, or Geriatric patients (patients aged 65 and older) in participating centers in Lebanon
* Presence of pain or fever necessitating the administration of Paracetamol
* Absence of an Intravenous Line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale pain scores for conscious and cooperative patients | 60 minutes
  This outcome measures the decrease in pain scores between t0 (right before acetaminophen administration) and t60 minutes using the Numerical Rating Scale in conscious and cooperative patients, where 10/10 is the worst imaginable pain and 0/10 is no pain at all.
  A Minimal Clinically Important Difference (MCID) of 2/10 is set to define efficacy.
Change on Algoplus Pain Scale for patients with verbal communication difficulties | 60 minutes
  This outcome measures the decrease in pain scores between t0 (right before acetaminophen administration) and t60 minutes using Algoplus Scale, a behavioural rating scale for acute pain for patients with verbal communication difficulties. A score of 2 or above diagnoses pain with 87% sensitivity and 80% specificity.
  The scale evaluates facial expressions, look, complaints, body position and atypical behaviours of patients with verbal communication difficulties.
  Each item marked "yes" is awarded one point and the total across all the items gives a total score out of 5.
  Efficacy is defined as a decrease of the score to less than 2/5.
Change in temperature measurement | 60 minutes
  Decrease in temperature measurement. A Minimal Clinically Important Difference (MCID) of 0.5 degrees Celsius is set to define efficacy.
Appearance of local side effects | at the time of perfusion, after 30 minutes, 60 minutes and 180 minutes, and one day after line removal
  Any local side effect is reported, including:
  * edema,
  * induration,
  * erythema,
  * tenderness,
  * warmth,
  * abcess,
  * necrosis

SECONDARY OUTCOMES:
Early effect on pain in conscious and cooperative patients | 30 minutes
  To evaluate if any early effect on pain is measurable, this outcome measures the pain scores at t30 minutes using the Numerical Rating Scale in conscious and cooperative patients, where 10/10 is the worst imaginable pain and 0/10 is no pain at all.
Sustained effect on pain in conscious and cooperative patients | 180 minutes
  To evaluate if the effect on pain is sustained over time, this outcome measures the pain scores at t180 minutes using the Numerical Rating Scale in conscious and cooperative patients, where 10/10 is the worst imaginable pain and 0/10 is no pain at all.
Early effect on pain in patients with verbal communication difficulties | 30 minutes
  To evaluate if any early effect on pain is measurable, this outcome measures the pain scores at t60 minutes and t180 minutes using Algoplus Scale, a behavioural rating scale for acute pain for patients with verbal communication difficulties. A score of 2 or above diagnoses pain with 87% sensitivity and 80% specificity.
  The scale evaluates facial expressions, look, complaints, body position and atypical behaviours of patients with verbal communication difficulties.
  Each item marked "yes" is awarded one point and the total across all the items gives a total score out of 5.
Sustained effect on pain in patients with verbal communication difficulties | 180 minutes
  To evaluate if the effect on pain is sustained over time, this outcome measures the pain scores at t180 minutes using Algoplus Scale, a behavioural rating scale for acute pain for patients with verbal communication difficulties. A score of 2 or above diagnoses pain with 87% sensitivity and 80% specificity.
  The scale evaluates facial expressions, look, complaints, body position and atypical behaviours of patients with verbal communication difficulties.
  Each item marked "yes" is awarded one point and the total across all the items gives a total score out of 5.
Early effect on fever | 30 minutes
  To evaluate if any early effect on fever is measurable, temperature is measured at t30 minutes.
Sustained effect on fever | 180 minutes
  To evaluate if the effect on fever is sustained over time, temperature is measured at t180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joe El Khoury, MD, Principal Investigator — Hotel-Dieu de France
Locations (1):
- Hotel-Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No